CLINICAL TRIAL: NCT01303159
Title: Pilot Study to Assess Safety and Efficacy of an Endoscopic Bipolar Radiofrequency Probe (ENDOHPB) in the Management of Unresectable Bile Duct and Pancreatic Cancer
Brief Title: Endoscopic Bipolar Radiofrequency Probe (ENDOHPB) in the Management of Unresectable Bile Duct and Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: EndoHPB probe is FDA approved and considered standard of care
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: EMcision Limited (Unknown)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1107011793
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Cholangiocarcinoma; Pancreatic Cancer
Keywords: Cholangiocarcinoma; Pancreatic Cancer; Radiofrequency; Ablation
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiofrequency probe (ENDOHPB) (Experimental): Intervention:
  The EndoHPB is an endoscopic bipolar catheter designed to ablate tissue in malignant tumors within luminal structures, such as the biliary tree or pancreatic ducts. EndoHPB can be deployed via an ERCP or Percutaneous Transhepatic Cholangiographic (PTC) route. By using radiofrequency (RF) energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may delay tumour growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent deployment
  Interventions: Device: Endoscopic bipolar radiofrequency probe (ENDOHPB)

INTERVENTIONS:
Device: Endoscopic bipolar radiofrequency probe (ENDOHPB) — EndoHPB (EMcision Ltd, UK) is a single use sterile device for use at ERCP or PTC. It is a 8F (2.6mm) catheter with a 1.8m working length, that is designed to be inserted into the target duct of the hepatic, biliary or pancreatic system over a guide wire. The device is compatible with endoscopes that have a working channel of 3.2mm or greater. It comprises of a coaxial over the wire (OTW) catheter with 2 ring electrodes spaced 8mm apart at its distal end. The distal electrode is 5mm from the leading edge of the catheter. The two electrodes at the distal end of EndoHPB are designed to produce a heating zone length of approximately 25 mm.
  Other Names: EndoHPB (EMcision Ltd, UK)

SUMMARY:
The purpose of this study is to assess safety and ability of the endoscopic bipolar radiofrequency ablation (RFA) probe (ENDOHPB) to produce an improvement in the management of cancer of the bile duct or the pancreatic duct. By using radiofrequency (RF) energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may delay tumour growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent deployment. The study will look to see if the ENDOHPB is able to keep the stent open longer and perhaps decrease the number of invasive procedures for occluded (blocked) stents.

DETAILED DESCRIPTION:
Only a small proportion of patients with biliary obstruction caused by cholangiocarcinoma or pancreatic cancer are suitable for surgical resection. As the cancer grows, it blocks the drainage of the bile ducts that carry digestive juices from the gall bladder and pancreas to the small intestine. Blocked drainage causes abdominal pain, bloating, and nausea. ERCP (endoscopic retrograde cholangiopancreatography) is often prescribed. ERCP with stent placement is the standard medical procedure for people with bile duct and pancreatic cancer.

The purpose of this study is to assess safety and ability of the endoscopic bipolar radiofrequency ablation (RFA) probe (ENDOHPB) to produce an improvement in the management of cancer of the bile duct or the pancreatic duct. By using radiofrequency (RF) energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may delay tumour growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent deployment. The study will look to see if the ENDOHPB is able to keep the stent open longer and perhaps decrease the number of invasive procedures for occluded (blocked) stents.

The objectives are:

• To assess assess the safety and effectiveness of an endoscopic bipolar radiofrequency catheter (EndoHPB) in the management of unresectable cholangiocarcinoma and pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Either gender greater than or equal to 18 years of age.
* Pancreatic cancer or cholangiocarcinoma unsuitable for surgical resection. Criteria of unresectability being based on 1) metastatic disease or 2) locally advanced.
* Biliary obstruction
* Blocked self expanding mesh metal stent (SEMS)
* Subjects capable of giving informed consent
* Life expectancy of at least 3 months

Exclusion Criteria:

* Cardiac Pacemaker
* Patient unstable for endoscopy
* Inability to give informed consent
* Uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01-13 (Actual); Study Completion 2014-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Result] Figueroa-Barojas P, Bakhru MR, Habib NA, Ellen K, Millman J, Jamal-Kabani A, Gaidhane M, Kahaleh M. Safety and efficacy of radiofrequency ablation in the management of unresectable bile duct and pancreatic cancer: a novel palliation technique. J Oncol. 2013;2013:910897. doi: 10.1155/2013/910897. Epub 2013 Apr 8. PMID 23690775

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiofrequency Probe (ENDOHPB): Intervention:
  The EndoHPB Radiofrequency probe
Period: Overall Study
Arm/Group | Radiofrequency Probe (ENDOHPB)
Started | 29
Completed | 6
Not Completed | 23
Not completed — Death | 16
Not completed — Study Termination | 7

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Probe (ENDOHPB)
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bile Duct Stricture Diameter
Description: To assess effectiveness of an endoscopic bipolar radiofrequency catheter (EndoHPB) in the management of unresectable cholangiocarcinoma and pancreatic cancer
Time Frame: 2 years
Population: Participants not analyzed has study was terminated before follow up data could be collected.
Arm/Group | Radiofrequency Probe (ENDOHPB)
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: To assess safety of an endoscopic bipolar radiofrequency catheter (EndoHPB) in the management of unresectable cholangiocarcinoma and pancreatic cancer
Time Frame: 2 years
Population: Preliminary analyses because study was terminated before follow up data could be collected.
Measure: Number; unit: participants
Arm/Group | Radiofrequency Probe (ENDOHPB)
Number analyzed (Participants) | 29
participants | 16

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Radiofrequency Probe (ENDOHPB)
All-Cause Mortality (participants affected / at risk) | 16/29
Serious Adverse Events (participants affected / at risk) | 16/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Probe (ENDOHPB) (N=29)
Fever (Gastrointestinal disorders) | 4 (4)
Death (Gastrointestinal disorders) | 16 (16)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early study termination leading to no preliminary analyses. Total enrolled 29, only 6 subjects had follow up data of 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No